CLINICAL TRIAL: NCT04494477
Title: The Evaluation of IN•Clued - Inclusive Health Care: Youth & Providers Empowered
Brief Title: Evaluation of the Impact of the IN•Clued Curriculum: An LGBTQ Sex ed Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philliber Research & Evaluation (Other)
Collaborators: Planned Parenthood of the Great Northwest and Hawaiian Islands (Other); The Office of Adolescent Health, HHS (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ashley Philliber, Principal Investigator, Philliber Research & Evaluation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PhilliberINclued
Record Dates: First submitted 2020-07-22; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Teen Pregnancy; STD Prevention
Keywords: LGBTQ sex education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The IN•clued program (Experimental): The IN•clued program for youth consists of a three-hour in-person workshop for youth which includes lessons about safe sex practices and self-efficacy at healthcare centers, exam room roleplays, and a discussion on patient rights. Youth receive a Zine, or a magazine-style booklet, that they may take home. They also receive a list of local healthcare providers that highlights those that have participated in the IN•clued healthcare provider workshop or have had training on working with the LGBTQ population. Program youth can also receive text messages with health tips and reminders to visit a healthcare center.
  Interventions: Behavioral: The IN•clued program
- Control (No Intervention): The youth control group receives a 10-minute presentation and a list of local sexual healthcare providers, with no indication of which providers have been trained to be more LGBTQ friendly and accepting. This 10-minute presentation is a part of a longer three-hour activity unrelated to sexual health or accessing sexual healthcare. During the three-hour session, the list of approved activities includes but is not limited to:
  * Films by, and for, LGBTQ youth about sexual orientation and gender identity;
  * Community scavenger hunts;
  * Poetry slams;
  * Discussions about relationships; and
  * Activities related to the appreciation of individuals' unique strengths.

INTERVENTIONS:
Behavioral: The IN•clued program — The INclued program as previously described.
  Arms: The IN•clued program

SUMMARY:
The INclued program was implemented in 16 states across the US. The purpose of this study is to measure: Nine months after the end of the program and one year after the workshop, are IN•clued participants less likely to report engaging in risky sexual behavior in the past three months compared to control group participants?

DETAILED DESCRIPTION:
The IN•clued program for youth consists of a three-hour in-person workshop for youth which includes lessons about safe sex practices and self-efficacy at healthcare centers, exam room roleplays, and a discussion on patient rights. Youth receive a Zine, or a magazine-style booklet, that they may take home. They also receive a list of local healthcare providers that highlights those that have participated in the IN•clued healthcare provider workshop or have had training on working with the LGBTQ population. Program youth can also receive text messages with health tips and reminders to visit a healthcare center.

Workshops take place with LGBTQ youth groups through schools, community-based organizations, or conferences. Each segment is led by adult facilitators or trained peer educators with adult facilitator support. These peer educators are from the Planned Parenthood Teen Council peer education program. Teen Council is a unique peer education program created in 1989 by PPGNHI. It is a strong and successful peer education program that trains high school youth to become experts in delivering inclusive, comprehensive sexual health education to their peers via group and community presentations. If trained peer educators are used, they implement the intervention with the guidance and oversight of an adult facilitator.

Participants in the control condition receive a benign intervention, which like IN•clued, meets in a group setting.

Once a site or group is defined, facilitators send implementation forms to Philliber. The evaluation team reviews the information and asks any needed questions which vary by group or site. The two groups cannot differ in any significant way (e.g., gender, SES, ethnicity, or special characteristic such as pregnant and parenting participants). All decisions about final eligibility are made by the research team. If two groups or sites are similar, they are approved. If they differ in a significant way, they are not eligible for the study.

Random assignment of the groups does not technically occur until the baseline administration of the survey is completed as participants can be both added and subtracted from the group list until the time of survey administration. One facilitator at each location is informed of the outcome of random assignment before or during the administration of the baseline survey. This is done so random assignment can occur immediately after surveys are conducted as this is a one-time workshop and participants do not give assent to participate until this time.

ELIGIBILITY:
Inclusion Criteria:

* Youth participants are already in LGBTQ groups, such as gay-straight alliances in schools or local community groups or those who are recruited to attend a special event at a community-based organization or conference. Participants must be at least 14 and preferably younger than 20. Ideally, they are part of the LGBTQ community, although this is not required.

Exclusion Criteria:

* Cannot require ESL support.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1401 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Nine months after the end of the program are IN•clued participants less likely to report engaging in risky sexual behavior in the past three months compared to control group participants? | One year after baseline
  If participants had recent (in the past three months) vaginal sex without a condom or birth control, recent oral sex without protection, or recent anal sex without a condom, they were coded as having engaged in recent unprotected or risky sexual behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Ash Philliber, PhD, Principal Investigator — Philliber Research & Evaluation
Locations (1):
- Philliber Research & Evaluation, Accord, New York, United States

REFERENCES:
- [Derived] Philliber A. The IN.clued Program: A Randomized Control Trial of an Effective Sex Education Program for Lesbian, Gay, Bisexual, Transgender, Queer, and Questioning Youths. J Adolesc Health. 2021 Oct;69(4):636-643. doi: 10.1016/j.jadohealth.2021.04.002. Epub 2021 May 14. PMID 33994311